CLINICAL TRIAL: NCT04731922
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TAK-510 in Healthy Subjects
Brief Title: A Study of TAK-510 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: TAK-510-1001; U1111-1261-6974 (Registry Identifier: WHO)
Record Dates: First submitted 2021-01-27; First posted 2021-02-01 (Actual); Results first posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2023-07

CONDITIONS: Healthy Participants
Keywords: Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TAK-510: Part 1 (Experimental): TAK-510 at starting dose of 5 microgram (mcg) or placebo-matching solution, subcutaneously, once on Day 1. Staggered dosing will be done in the first cohort of Part A (Cohort 1). Staggered dosing in subsequent Cohorts (Cohorts 2-12 and 21-25) will be used based on emerging safety, tolerability, and PK data from Cohort 1 as determined in the dose escalation meeting.
  Interventions: Drug: TAK-510; Drug: TAK-510 Placebo
- TAK-510: Part 2 (Experimental): TAK-510 to be decided (TBD) or placebo-matching solution, subcutaneously, once daily from Day 1 through Day 5. Dose of MRD Cohorts (Cohorts 13-17 and 26-28) of Part 2 will be determined based on emerging safety, tolerability, and available PK data from Part 1 (SRD) and any available PK data from Part 2 as determined in the dose escalation meeting.
  Interventions: Drug: TAK-510; Drug: TAK-510 Placebo
- TAK-510: Part 3 (Experimental): TAK-510 TBD or placebo-matching solution, subcutaneously, once daily from Days 1 to 7. Dose of dose titration and redosing Cohorts (Cohorts 18-20) of Part 3 will be based on emerging safety, tolerability, and available PK data from Part 1 (SRD) and Part 2 (MRD) as determined in the dose escalation meeting. Single redosing will be performed on Day 14 after 7 days of washout period following the 7 days treatment period.
  Interventions: Drug: TAK-510; Drug: TAK-510 Placebo

INTERVENTIONS:
Drug: TAK-510 — TAK-510 solution.
Drug: TAK-510 Placebo — TAK-510 placebo-matching solution.

SUMMARY:
This is a study of TAK-510 for people with symptoms of feeling sick (nausea) or being sick (vomiting).

The main aims of the study are to check if healthy adults have side effects from TAK-510 and to check how much TAK-510 they can receive without getting side effects from it.

The study will be in 3 parts. Participants will take part in only 1 of the 3 parts of the study.

At the first visit, the study doctor will check if each person can take part. For those who can take part, they will be placed in 1 of many small groups. The 1st groups will join Part 1 of the study, the 2nd groups will join Part 2 and the 3rd groups will join Part 3. They will receive an injection under the skin of either TAK-510 or placebo. In this study, a placebo will look like the TAK-510 injection but will not have any medicine in it.

In Part 1, the 1st group of participants will receive 1 injection of either TAK-510 or placebo. Different participants within this group will receive lower to higher doses of TAK-510. The participants in this group will stay in the clinic for 4 days after their injection for some tests and check for any side effects from their treatment.

In Part 2, the 2nd group of participants will receive an injection of either TAK-510 or placebo, once a day for 5 days. Different participants within this group will receive lower to higher doses of TAK-510. The participants in this group will stay in the clinic for 9 days after their 1st injection for some tests and check for any side effects from their treatment.

In Part 3, the 3rd group of participants will visit the clinic 2 times. At the 1st visit, they will receive an injection either of TAK-510 or placebo, once a day for 7 days. Each participant in this group will receive lower to higher doses of TAK-510. They will stay in the clinic for 8 days after their 1st injection for some tests and check for any side effects from their treatment.

At the 2nd clinic visit, each participant will receive 1 single injection of TAK-510 or placebo. This will happen 7 days after their last injection from the previous clinic visit. They will receive the same dose as their previous dose. They will stay in the clinic for 3 days for some tests and check for any side effects from their treatment.

After treatment, all participants in the study will return to the clinic for a weekly check-up visit for up to 3 weeks.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-510. The study will look at the safety, tolerability, and PK of TAK-510 in healthy participants.

The study will enroll up to approximately 224 healthy participants. Participants in each cohort will be randomized to receive treatment with TAK-510 or matching placebo which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need). The study consists of 3 parts and up to 28 cohorts as mentioned below.

* TAK-510, Part 1: Single rising dose (SRD) design to assess the safety, immunogenicity, tolerability, and PK of TAK-510
* TAK-510, Part 2: Multiple rising dose (MRD) design to assess the safety, immunogenicity, tolerability, and PK of TAK-510
* TAK-510, Part 3: Dose titration and redosing design to assess the safety, immunogenicity, tolerability, and PK of TAK-510

This multi-center trial will be conducted in the United States. The overall duration of the study is approximately 57 days. Participants will be followed up for 7 days after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Continuous nonsmoker who has not used nicotine- and tobacco-containing products for at least 3 months prior to dosing and throughout the study.
* Body mass index (BMI) greater than or equal to (>=) 18.0 and less than or equal to (<=) 30.0 kilogram per square meter (kg/m^2) at the screening visit.

Exclusion Criteria:

* Has a positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency antibody/antigen, at the screening visit.
* Had major surgery or donated or lost 1 unit of blood (approximately 500 milliliter [mL]) within 4 weeks before the screening visit.
* Unable to refrain from or anticipates using all medications including herbal medicines beginning approximately 7 days before administration of the first dose of study drug, throughout the study until 2 days after discharge.
* Unable to refrain from or anticipates using marijuana or cannabis-containing products beginning approximately 7 days before administration of the first dose of study drug, throughout the study until after the last PK dose.
* Has had a previous major psychotic disorder.
* Has an average semirecumbent blood pressure (BP) less than 90/60 millimeter of mercury (mmHg) or greater than 140/90 mmHg from screening to predose, inclusive. Any assessments on Day -1, where 2 consecutive time point values do not meet this criterion must be discussed with the medical monitor for approval.
* Has orthostatic hypotension defined as a decrease in systolic BP >=20 mmHg or a decrease in diastolic BP >=10 mmHg at approximately 3 minutes of standing when compared with BP from the semirecumbent position, at screening to predose assessments, inclusive. In asymptomatic participants, any assessments after screening that do not meet this criterion may be repeated after the participant has remained in the semirecumbent or supine position for 15 minutes. If the repeat assessment is exclusionary based on the above criterion, the participant will not be eligible. If the repeat assessment is not exclusionary, the participant will be eligible.
* Has postural orthostatic tachycardia, defined as an increase of greater than (>) 30 beats per minute (bpm) or heart rate (HR) >120 bpm at approximately 3 minutes, of standing, at screening to predose assessments, inclusive. Any assessments after screening that do not meet this criterion may be repeated with the participant remaining standing for up to a total of 5 minutes, provided that the participant remains asymptomatic. If the repeat assessment occurring within 5 minutes is exclusionary based on the above criterion, the participant will not be eligible. A confirmed orthostatic increase of >30 bpm, but less than (<) 40 bpm, on 1 or more Day -1 assessments may not be considered exclusionary if not considered clinically significant by the investigator and the medical monitor. Such assessments must be discussed with the medical monitor prior to determination that the participant is eligible to proceed.
* Has a known or suspected current coronavirus disease 2019 (COVID-19) infection or is at risk of COVID-19 infection as assessed by the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2022-07-24 (Actual); Study Completion 2022-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (2):
- United States (2):
  - PPD Development, LP, Las Vegas, Nevada
  - PPD Development, LP, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click on this link — https://clinicaltrials.takeda.com/study-detail/602005c75f53e3001ed0d7bc

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in the United States from 3 February 2021 to 24 July 2022.
Pre-assignment Details: Healthy participants were enrolled in study into 2 Parts: Single Rising Doses (SRD) (Part 1) and Multiple Rising Doses (MRD) (Part 2) to receive TAK-510 placebo-matching or TAK-510 injection. Starting Dose 1 was 5 micrograms (mcg) and subsequent doses were increased from low dose to high dose for Doses 1-11 and Doses 1A-4A in Part 1 or Part 2, respectively. Study was completed after completion of Parts 1 and 2. Sponsor decided not to conduct Part 3 after comprehensive review of available data.
Groups:
- Part 1, SRD Cohorts 1 to 11: Pooled Placebo: TAK-510 placebo-matching injection, subcutaneously, once on Day 1.
- Part 1, SRD Cohort 1: TAK-510 Dose 1: TAK-510 Dose 1, injection, subcutaneously, once on Day 1.
- Part 1, SRD Cohort 2: TAK-510 Dose 2: TAK-510 Dose 2, injection, subcutaneously, once on Day 1. The dose of TAK-510 was based on 24-hours safety, tolerability, laboratory results and available pharmacokinetic (PK) data from previous SRD Cohort 1.
- Part 1, SRD Cohort 3: TAK-510 Dose 3: TAK-510 Dose 3, injection, subcutaneously, once on Day 1. The dose of TAK-510 was based on 24-hours safety, tolerability, laboratory results and available PK data from previous SRD Cohort.
- Part 1, SRD Cohort 4: TAK-510 Dose 4: TAK-510 Dose 4, injection, subcutaneously, once on Day 1. The dose of TAK-510 was based on 24-hours safety, tolerability, laboratory results and available PK data from previous SRD Cohort.
- Part 1, SRD Cohort 5: TAK-510 Dose 5: TAK-510 Dose 5, injection, subcutaneously, once on Day 1. The dose of TAK-510 was based on 24-hours safety, tolerability, laboratory results and available PK data from previous SRD Cohort.
- Part 1, SRD Cohort 6: TAK-510 Dose 6: TAK-510 Dose 6, injection, subcutaneously, once on Day 1. The dose of TAK-510 was based on 24-hours safety, tolerability, laboratory results and available PK data from previous SRD Cohort.
- Part 1, SRD Cohort 7: TAK-510 Dose 7: TAK-510 Dose 7, injection, subcutaneously, once on Day 1. The dose of TAK-510 was based on 24-hours safety, tolerability, laboratory results and available PK data from previous SRD Cohort.
- Part 1, SRD Cohort 8: TAK-510 Dose 8: TAK-510 Dose 8, injection, subcutaneously, once on Day 1. The dose of TAK-510 was based on 24-hours safety, tolerability, laboratory results and available PK data from previous SRD Cohort.
- Part 1, SRD Cohort 9: TAK-510 Dose 9: TAK-510 Dose 9, injection, subcutaneously, once on Day 1. The dose of TAK-510 was based on 24-hours safety, tolerability, laboratory results and available PK data from previous SRD Cohort.
- Part 1, SRD Cohort 10: TAK-510 Dose 10: TAK-510 Dose 10, injection, subcutaneously, once on Day 1. The dose of TAK-510 was based on 24-hours safety, tolerability, laboratory results and available PK data from previous SRD Cohort.
- Part 1, SRD Cohort 11: TAK-510 Dose 11: TAK-510 Dose 11, injection, subcutaneously, once on Day 1. The dose of TAK-510 was based on 24-hours safety, tolerability, laboratory results and available PK data from previous SRD Cohort.
- Part 2, MRD 12 to 15 Cohorts: Pooled Placebo: TAK-510 placebo-matching placebo, injection, subcutaneously from Days 1 to 5.
- Part 2, MRD Cohort 12: Dose 1A: TAK-510 Dose 1A, injection, subcutaneously from Days 1 to 5. The dose of TAK-510 was based on safety, tolerability, and available PK data from SRD Part 1.
- Part 2, MRD Cohort 13: Dose 2A: TAK-510 Dose 2A, injection, subcutaneously from Days 1 to 5. The dose of TAK-510 was based on safety, tolerability, and available PK data from Part 1 and review of safety, tolerability, and available PK data from previous MRD Cohort.
- Part 2, MRD Cohort 14: Dose 3A: TAK-510 Dose 3A, injection, subcutaneously from Days 1 to 5. The dose of TAK-510 was based on safety, tolerability, and available PK data from Part 1 and review of safety, tolerability, and PK data from previous MRD Cohort.
- Part 2, MRD Cohort 15: Dose 4A: TAK-510 Dose 4A, injection, subcutaneously from Days 1 to 5. The dose of TAK-510 was based on safety, tolerability, and available PK data from Part 1 and review of safety, tolerability, and PK data from previous MRD Cohort.
Period: Overall Study
Arm/Group | Part 1, SRD Cohorts 1 to 11: Pooled Placebo | Part 1, SRD Cohort 1: TAK-510 Dose 1 | Part 1, SRD Cohort 2: TAK-510 Dose 2 | Part 1, SRD Cohort 3: TAK-510 Dose 3 | Part 1, SRD Cohort 4: TAK-510 Dose 4 | Part 1, SRD Cohort 5: TAK-510 Dose 5 | Part 1, SRD Cohort 6: TAK-510 Dose 6 | Part 1, SRD Cohort 7: TAK-510 Dose 7 | Part 1, SRD Cohort 8: TAK-510 Dose 8 | Part 1, SRD Cohort 9: TAK-510 Dose 9 | Part 1, SRD Cohort 10: TAK-510 Dose 10 | Part 1, SRD Cohort 11: TAK-510 Dose 11 | Part 2, MRD 12 to 15 Cohorts: Pooled Placebo | Part 2, MRD Cohort 12: Dose 1A | Part 2, MRD Cohort 13: Dose 2A | Part 2, MRD Cohort 14: Dose 3A | Part 2, MRD Cohort 15: Dose 4A
Started | 23 | 6 | 6 | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 6 | 6 | 6
Completed | 22 | 6 | 6 | 5 | 6 | 5 | 4 | 6 | 6 | 6 | 5 | 6 | 8 | 7 | 6 | 6 | 6
Not Completed | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study treatment.
Groups:
- Part 1, SRD Cohort 2: TAK-510 Dose 2: TAK-510 Dose 2, injection, subcutaneously, once on Day 1. The dose of TAK-510 was based on 24-hours safety, tolerability, laboratory results and available PK data from previous SRD Cohort 1.
- Total: Total of all reporting groups
Arm/Group | Part 1, SRD Cohorts 1 to 11: Pooled Placebo | Part 1, SRD Cohort 1: TAK-510 Dose 1 | Part 1, SRD Cohort 2: TAK-510 Dose 2 | Part 1, SRD Cohort 3: TAK-510 Dose 3 | Part 1, SRD Cohort 4: TAK-510 Dose 4 | Part 1, SRD Cohort 5: TAK-510 Dose 5 | Part 1, SRD Cohort 6: TAK-510 Dose 6 | Part 1, SRD Cohort 7: TAK-510 Dose 7 | Part 1, SRD Cohort 8: TAK-510 Dose 8 | Part 1, SRD Cohort 9: TAK-510 Dose 9 | Part 1, SRD Cohort 10: TAK-510 Dose 10 | Part 1, SRD Cohort 11: TAK-510 Dose 11 | Part 2, MRD 12 to 15 Cohorts: Pooled Placebo | Part 2, MRD Cohort 12: Dose 1A | Part 2, MRD Cohort 13: Dose 2A | Part 2, MRD Cohort 14: Dose 3A | Part 2, MRD Cohort 15: Dose 4A | Total
Number analyzed (Participants) | 23 | 6 | 6 | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 6 | 6 | 6 | 124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 6 | 6 | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 6 | 6 | 6 | 124
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 17
  Male | 17 | 3 | 5 | 6 | 7 | 5 | 5 | 6 | 6 | 5 | 6 | 5 | 8 | 6 | 6 | 5 | 6 | 107
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 3 | 1 | 1 | 1 | 1 | 4 | 3 | 0 | 0 | 3 | 4 | 3 | 1 | 1 | 1 | 34
  Not Hispanic or Latino | 18 | 4 | 3 | 5 | 6 | 5 | 5 | 2 | 3 | 6 | 6 | 3 | 4 | 5 | 5 | 5 | 5 | 90
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 2 | 0 | 1 | 1 | 1 | 2 | 1 | 16
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Black or African American | 6 | 1 | 3 | 3 | 6 | 2 | 3 | 1 | 3 | 3 | 0 | 3 | 2 | 2 | 4 | 3 | 3 | 48
  White | 12 | 4 | 3 | 2 | 0 | 3 | 1 | 4 | 1 | 1 | 4 | 3 | 4 | 5 | 1 | 1 | 2 | 51
  More than one race | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 6 | 6 | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 6 | 6 | 6 | 124

OUTCOME MEASURES:

1. Primary Outcome: Parts 1 and 2: Number of Participants Who Met the Markedly Abnormal Criteria for Vital Sign Measurements at Least Once Post Dose
Description: Vital signs included systolic and diastolic blood pressure, body temperature, pulse rate (PR), respiratory rate, orthostatic blood pressure and pulse rate assessments. The markedly abnormal value (MAV) criteria for vital signs were systolic blood pressure (SBP) less than (<) 85 millimeter of mercury (mmHg), greater than (>) 180 mmHg; diastolic blood pressure (DBP) <50 mmHg, >110 mmHg; body temperature <35.6 degree Celsius, >37.7 degree Celsius; PR <50 beats per minute (bpm), >120 bpm; respiratory rate <12 breaths per minute (breaths/minute), >16 breaths/minute; orthostatic hypotension decrease in SBP greater than or equal to (>=) 20 mmHg or a decrease in DBP >=10 mmHg on standing; orthostatic tachycardia defined as an increase of >30 bpm or heart rate (HR) >120 bpm on standing. Number of participants who met the MAV criteria for vital signs at least once post dose were reported.
Time Frame: Parts 1 and 2: From the first dose of study drug up to Day 29
Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, SRD Cohorts 1 to 11: Pooled Placebo | Part 1, SRD Cohort 1: TAK-510 Dose 1 | Part 1, SRD Cohort 2: TAK-510 Dose 2 | Part 1, SRD Cohort 3: TAK-510 Dose 3 | Part 1, SRD Cohort 4: TAK-510 Dose 4 | Part 1, SRD Cohort 5: TAK-510 Dose 5 | Part 1, SRD Cohort 6: TAK-510 Dose 6 | Part 1, SRD Cohort 7: TAK-510 Dose 7 | Part 1, SRD Cohort 8: TAK-510 Dose 8 | Part 1, SRD Cohort 9: TAK-510 Dose 9 | Part 1, SRD Cohort 10: TAK-510 Dose 10 | Part 1, SRD Cohort 11: TAK-510 Dose 11 | Part 2, MRD 12 to 15 Cohorts: Pooled Placebo | Part 2, MRD Cohort 12: Dose 1A | Part 2, MRD Cohort 13: Dose 2A | Part 2, MRD Cohort 14: Dose 3A | Part 2, MRD Cohort 15: Dose 4A
Number analyzed (Participants) | 23 | 6 | 6 | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 6 | 6 | 6
Participants
  Temperature, <35.6 Degree Celsius | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Temperature, >37.7 Degree Celsius | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SBP, Standing: <85 mmHg | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  SBP, Standing: >180 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DBP, Standing: <50 mmHg | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3
  DBP, Standing: >110 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR, Standing: <50 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR, Standing: >120 bpm | 0 | 0 | 0 | 1 | 2 | 4 | 2 | 2 | 5 | 4 | 5 | 2 | 1 | 4 | 1 | 4 | 4
  SBP, Semi-Recumbent: <85 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SBP, Semi-Recumbent: >180 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DBP, Semi-Recumbent: <50 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  DBP, Semi-Recumbent: >110 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR, Semi-Recumbent: <50 bpm | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR, Semi-Recumbent: >120 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Respiratory Rate, Semi-Recumbent: <12 breaths/minute | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 4 | 4 | 5 | 0 | 1
  Respiratory Rate, Semi-Recumbent: >16 breaths/minute | 10 | 4 | 3 | 3 | 2 | 3 | 5 | 1 | 3 | 3 | 3 | 2 | 6 | 4 | 4 | 5 | 5
  Orthostatic SBP: Decrease in SBP >=20 mmHg on standing | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3
  Orthostatic DBP: Decrease in DBP >=10 mmHg on standing | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Orthostatic PR: Increase of >30 or HR >120 mmHg on standing | 6 | 0 | 3 | 3 | 3 | 5 | 2 | 4 | 6 | 4 | 6 | 2 | 4 | 6 | 3 | 6 | 5

2. Primary Outcome: Parts 1 and 2: Number of Participants Who Met the Markedly Abnormal Criteria for Electrocardiogram (ECG) Parameters at Least Once Post Dose
Description: ECG included HR, PR, QT interval with Fridericia correction (QTcF) interval and QRS duration. The MAV criteria for 12-lead ECG parameters included heart rate <50 bpm, >120 bpm; PR interval less than or equal to (<=)80 milliseconds (msec), >=200 msec; QTcF interval >=500 msec; QRS duration <=80 msec, >=120 msec. Number of participants who met the MAV criteria for ECG parameters at least once post dose were reported.
Time Frame: Parts 1 and 2: From the first dose of study drug up to Day 29
Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, SRD Cohorts 1 to 11: Pooled Placebo | Part 1, SRD Cohort 1: TAK-510 Dose 1 | Part 1, SRD Cohort 2: TAK-510 Dose 2 | Part 1, SRD Cohort 3: TAK-510 Dose 3 | Part 1, SRD Cohort 4: TAK-510 Dose 4 | Part 1, SRD Cohort 5: TAK-510 Dose 5 | Part 1, SRD Cohort 6: TAK-510 Dose 6 | Part 1, SRD Cohort 7: TAK-510 Dose 7 | Part 1, SRD Cohort 8: TAK-510 Dose 8 | Part 1, SRD Cohort 9: TAK-510 Dose 9 | Part 1, SRD Cohort 10: TAK-510 Dose 10 | Part 1, SRD Cohort 11: TAK-510 Dose 11 | Part 2, MRD 12 to 15 Cohorts: Pooled Placebo | Part 2, MRD Cohort 12: Dose 1A | Part 2, MRD Cohort 13: Dose 2A | Part 2, MRD Cohort 14: Dose 3A | Part 2, MRD Cohort 15: Dose 4A
Number analyzed (Participants) | 23 | 6 | 6 | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 6 | 6 | 6
Participants
  ECG HR, <50 bpm | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ECG HR, >120 bpm | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 1
  PR Interval, <=80 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  PR Interval, >=200 msec | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
  QRS Duration, <=80 msec | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
  QRS Duration, >=120 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  QTcF Interval, >=500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

3. Primary Outcome: Parts 1 and 2: Number of Participants Who Met the Markedly Abnormal Criteria for Laboratory Value at Least Once Post Dose
Description: Clinical laboratory parameters included tests for chemistry and hematology. The MAV criteria for laboratory value included hemoglobin <0.8*LLN,>1.2*ULN; hematocrit <0.8*LLN,>1.2*ULN;RBC count <0.8*LLN, >1.2*ULN;WBC count <0.5*LLN, >1.5*ULN; platelet count <75*10^9 per liter, >600*10^9 per liter; ALT >3*ULN; AST >3*ULN,GGT >3*ULN, normal baseline; >2*baseline,abnormal baseline; ALP>3*ULN, normal baseline; >2*baseline, abnormal baseline; total bilirubin >1.5*ULN, normal baseline; >1.5* baseline, abnormal baseline; albumin <25g/L; total protein <0.8* LLN, >1.2*ULN; creatinine >177 micromole per liter; blood urea nitrogen >10.7 mmol/L; sodium <130 mmol/L, >150mmol/L; potassium <3.0mmol/L, >5.5 mmol/L; glucose <3mmol/L, >10mmol/L; chloride <75mmol/L, >126mmol/L; calcium corrected serum calcium of <LLN-8.0 mg/dL; <LLN-2.0mmol/L; ionized calcium <LLN-1.0mmol/L; bicarbonate <8.0mmol/L. Number of participants who met the MAV criteria for laboratory value at least once post dose were reported.
Time Frame: Parts 1 and 2: From the first dose of study drug up to Day 29
Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study treatment. Here, LLN = lower limit of normal; RBC = red blood cell; WBC = white blood cell; ALP = alkaline phosphatase; GGT = Gamma-glutamyl transferase; g/L = gram per liter; mmol/L = millimoles per liter; mg/dL = milligrams per deciliter.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1, SRD Cohort 5: TAK-510 Dose 5: TAK-510 Dose 5 injection, subcutaneously, once on Day 1. The dose of TAK-510 was based on 24-hours safety, tolerability, laboratory results and available PK data from previous SRD Cohort.
Arm/Group | Part 1, SRD Cohorts 1 to 11: Pooled Placebo | Part 1, SRD Cohort 1: TAK-510 Dose 1 | Part 1, SRD Cohort 2: TAK-510 Dose 2 | Part 1, SRD Cohort 3: TAK-510 Dose 3 | Part 1, SRD Cohort 4: TAK-510 Dose 4 | Part 1, SRD Cohort 5: TAK-510 Dose 5 | Part 1, SRD Cohort 6: TAK-510 Dose 6 | Part 1, SRD Cohort 7: TAK-510 Dose 7 | Part 1, SRD Cohort 8: TAK-510 Dose 8 | Part 1, SRD Cohort 9: TAK-510 Dose 9 | Part 1, SRD Cohort 10: TAK-510 Dose 10 | Part 1, SRD Cohort 11: TAK-510 Dose 11 | Part 2, MRD 12 to 15 Cohorts: Pooled Placebo | Part 2, MRD Cohort 12: Dose 1A | Part 2, MRD Cohort 13: Dose 2A | Part 2, MRD Cohort 14: Dose 3A | Part 2, MRD Cohort 15: Dose 4A
Number analyzed (Participants) | 23 | 6 | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 6 | 6 | 6
Participants
  Chemistry, Alanine Aminotransferase (ALT) (units per liter [U/L]: >3* upper limit of normal (ULN) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chemistry, Aspartate Aminotransferase (AST) (U/L): >3*ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0

4. Primary Outcome: Parts 1 and 2: Number of Participants Reporting One or More Treatment-emergent Adverse Event (TEAE)
Description: A TEAE was defined as an adverse event (AE) that started or worsened after first dose of the study treatment and within 30 days of last dose of study treatment. An AE was defined as any untoward medical occurrence in a clinical investigation participant who has signed informed consent to participate in a study; it did not necessarily had to have a causal relationship with the treatment. An AE could therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it was considered related to the drug.
Time Frame: From the first dose of study drug until 30 days after last dose in Parts 1 and 2 (SRD Cohorts: up to Day 31, MRD Cohorts: up to Day 35)
Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1, SRD Cohort 8: TAK-510 Dose 8: TAK-510 Dose 8 injection, subcutaneously, once on Day 1. The dose of TAK-510 was based on 24-hours safety, tolerability, laboratory results and available PK data from previous SRD Cohort.
Arm/Group | Part 1, SRD Cohorts 1 to 11: Pooled Placebo | Part 1, SRD Cohort 1: TAK-510 Dose 1 | Part 1, SRD Cohort 2: TAK-510 Dose 2 | Part 1, SRD Cohort 3: TAK-510 Dose 3 | Part 1, SRD Cohort 4: TAK-510 Dose 4 | Part 1, SRD Cohort 5: TAK-510 Dose 5 | Part 1, SRD Cohort 6: TAK-510 Dose 6 | Part 1, SRD Cohort 7: TAK-510 Dose 7 | Part 1, SRD Cohort 8: TAK-510 Dose 8 | Part 1, SRD Cohort 9: TAK-510 Dose 9 | Part 1, SRD Cohort 10: TAK-510 Dose 10 | Part 1, SRD Cohort 11: TAK-510 Dose 11 | Part 2, MRD 12 to 15 Cohorts: Pooled Placebo | Part 2, MRD Cohort 12: Dose 1A | Part 2, MRD Cohort 13: Dose 2A | Part 2, MRD Cohort 14: Dose 3A | Part 2, MRD Cohort 15: Dose 4A
Number analyzed (Participants) | 23 | 6 | 6 | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 6 | 6 | 6
Participants | 10 | 1 | 3 | 3 | 4 | 6 | 6 | 4 | 6 | 4 | 6 | 6 | 5 | 7 | 3 | 6 | 5

5. Secondary Outcome: Part 3, Number of Participants Who Met the Markedly Abnormal Criteria for Vital Sign Measurements at Least Once Post Single Subcutaneous Rechallenge Doses After a Washout From Multiple Subcutaneous Dose Regimens
Description: Vital signs included systolic and diastolic blood pressure, body temperature, PR, respiratory rate, orthostatic blood pressure and pulse rate assessments. The MAV criteria for vital signs were systolic SBP < 85 mmHg, >180 mmHg; DBP <50 mmHg, >110 mmHg; body temperature <35.6 degree Celsius, >37.7 degree Celsius; PR <50 bpm, >120 bpm; respiratory rate <12 breaths/minute, >16 breaths/minute; orthostatic hypotension decrease in SBP >=20 mmHg or a decrease in DBP >=10 mmHg on standing; orthostatic tachycardia defined as an increase of >30 bpm or HR >120 bpm on standing. Sponsor decided not to conduct Part 3 after comprehensive review of available data. No participants were enrolled in Part 3 of the study. Hence, no data collection and assessment were done in Part 3.
Time Frame: Part 3: From the first dose of study drug up to Day 29
Population: No participants were enrolled in Part 3 of the study. Hence, no data collection and assessment were done in Part 3.
Reporting Status: Not Posted

6. Secondary Outcome: Part 3, Number of Participants Who Met the Markedly Abnormal Criteria for ECG Parameters at Least Once Post Single Subcutaneous Rechallenge Doses After a Washout From Multiple Subcutaneous Dose Regimens
Description: ECG included HR, PR, QT QTcF interval and QRS duration. The MAV criteria for 12-lead ECG parameters included heart rate <50 bpm, >120 bpm; PR interval <=80 msec, >=200 msec; QTcF interval >=500 msec or >=30 msec change from baseline and >=450 msec; QRS duration <=80 msec, >=120 msec. Sponsor decided not to conduct Part 3 after comprehensive review of available data. No participants were enrolled in Part 3 of the study. Hence, no data collection and assessment were done in Part 3.
Time Frame: Part 3: From the first dose of study drug up to Day 29
Reporting Status: Not Posted

7. Secondary Outcome: Part 3, Number of Participants Who Met the Markedly Abnormal Criteria for Laboratory Value at Least Once Post Single Subcutaneous Rechallenge Doses After a Washout From Multiple Subcutaneous Dose Regimens
Description: MAV criteria: hemoglobin <0.8*LLN,>1.2*ULN; hematocrit <0.8*LLN,>1.2*ULN;RBC count <0.8*LLN, >1.2*ULN;WBC count <0.5*LLN, >1.5*ULN; platelet count <75*10^9 per liter, >600*10^9 per liter; ALT >3*ULN; AST >3*ULN,GGT >3*ULN, normal baseline; >2*baseline,abnormal baseline; ALP>3*ULN, normal baseline; >2*baseline, abnormal baseline; total bilirubin >1.5*ULN, normal baseline; >1.5* baseline, abnormal baseline; albumin <25g/L; total protein <0.8* LLN, >1.2*ULN; creatinine >177 micromole per liter; blood urea nitrogen >10.7 mmol/L; sodium <130 mmol/L, >150mmol/L; potassium <3.0mmol/L, >5.5 mmol/L; glucose <3mmol/L, >10mmol/L; chloride <75mmol/L, >126mmol/L; calcium corrected serum calcium of <LLN-8.0 mg/dL; <LLN-2.0mmol/L; ionized calcium <LLN-1.0mmol/L; bicarbonate <8.0mmol/L. Sponsor decided not to conduct Part 3 after comprehensive review of available data. No participants were enrolled in Part 3. Hence, no data collection and assessment were done in Part 3.
Time Frame: Part 3: From the first dose of study drug up to Day 29
Reporting Status: Not Posted

8. Secondary Outcome: Part 3, Number of Participants Reporting One or More TEAE Post Single Subcutaneous Rechallenge Doses After a Washout From Multiple Subcutaneous Dose Regimens
Description: A TEAE was defined as an AE that started or worsened after first dose of the study treatment and within 30 days of last dose of study treatment. An AE was defined as any untoward medical occurrence in a clinical investigation participant who has signed informed consent to participate in a study; it did not necessarily had to have a causal relationship with the treatment. An AE could therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it was considered related to the drug. Sponsor decided not to conduct Part 3 after comprehensive review of available data. No participants were enrolled in Part 3 of the study. Hence, no data collection and assessment were done in Part 3.
Time Frame: Part 3: From the first dose of study drug until 30 days after last dose (up to Day 37)
Reporting Status: Not Posted

9. Secondary Outcome: Parts 1 and 2: Number of Participants Based on Antidrug Antibody (ADA) Status (Positive and Negative) in Serum
Description: A 3-tiered ADA testing strategy was used in this study. A sample was initially screened for ADA by the ADA screening assay. Any positive sample in the screening assay was considered a potential positive, which was confirmed for true positivity by the confirmatory assay. If a sample was confirmed as an ADA true positive, ADA titer was assessed. ADA positive was defined as participants who had confirmed positive ADA status in at least 1 postbaseline assessments. ADA negative was defined as participants who did not have a confirmed negative ADA status in any post-baseline assessment.
Time Frame: Parts 1 and 2: From the first dose of study drug up to Day 29
Population: The immunogenicity analysis set included all participants who received at least 1 dose of study treatment and had the baseline sample and at least 1 postbaseline sample.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, SRD Cohorts 1 to 11: Pooled Placebo | Part 1, SRD Cohort 1: TAK-510 Dose 1 | Part 1, SRD Cohort 2: TAK-510 Dose 2 | Part 1, SRD Cohort 3: TAK-510 Dose 3 | Part 1, SRD Cohort 4: TAK-510 Dose 4 | Part 1, SRD Cohort 5: TAK-510 Dose 5 | Part 1, SRD Cohort 6: TAK-510 Dose 6 | Part 1, SRD Cohort 7: TAK-510 Dose 7 | Part 1, SRD Cohort 8: TAK-510 Dose 8 | Part 1, SRD Cohort 9: TAK-510 Dose 9 | Part 1, SRD Cohort 10: TAK-510 Dose 10 | Part 1, SRD Cohort 11: TAK-510 Dose 11 | Part 2, MRD 12 to 15 Cohorts: Pooled Placebo | Part 2, MRD Cohort 12: Dose 1A | Part 2, MRD Cohort 13: Dose 2A | Part 2, MRD Cohort 14: Dose 3A | Part 2, MRD Cohort 15: Dose 4A
Number analyzed (Participants) | 23 | 6 | 6 | 6 | 7 | 6 | 5 | 6 | 6 | 6 | 5 | 6 | 8 | 6 | 6 | 6 | 6
Participants
  ADA Negative | 20 | 6 | 6 | 6 | 7 | 6 | 5 | 6 | 5 | 4 | 5 | 6 | 8 | 6 | 6 | 6 | 4
  ADA Positive | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2

10. Secondary Outcome: Part 3: Number of Participants Based on ADA Status (Positive and Negative) in Serum
Description: A 3-tiered ADA testing strategy was used in this study. A sample was initially screened for ADA by the ADA screening assay. Any positive sample in the screening assay was considered a potential positive, which was confirmed for true positivity by the confirmatory assay. If a sample was confirmed as an ADA true positive, ADA titer was assessed. ADA positive was defined as participants who had confirmed positive ADA status in at least 1 postbaseline assessments. ADA negative was defined as participants who did not have a confirmed negative ADA status in any post-baseline assessment. Sponsor decided not to conduct Part 3 after comprehensive review of available data. No participants were enrolled in Part 3 of the study. Hence, no data collection and assessment were done in Part 3.
Time Frame: Part 3: From the first dose of study drug up to Day 29
Reporting Status: Not Posted

11. Secondary Outcome: Parts 1 and 2: Number of ADA Positive Participants Based on Low or High ADA Titer
Description: The high ADA titer was defined as participant who has at least 1 post-baseline ADA titer >16 and low ADA titer was defined as participant whose postbaseline ADA titers are all <=16. The low or high ADA titer was assessed in ADA positive participants only.
Time Frame: Parts 1 and 2: From the first dose of study drug up to Day 29
Population: The immunogenicity analysis set included all participants who received at least 1 dose of study treatment and had the baseline sample and at least 1 postbaseline sample. Here "overall number of participants analyzed" signifies those participants who had positive ADA status in at least 1 postbaseline assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, SRD Cohorts 1 to 11: Pooled Placebo | Part 1, SRD Cohort 1: TAK-510 Dose 1 | Part 1, SRD Cohort 2: TAK-510 Dose 2 | Part 1, SRD Cohort 3: TAK-510 Dose 3 | Part 1, SRD Cohort 4: TAK-510 Dose 4 | Part 1, SRD Cohort 5: TAK-510 Dose 5 | Part 1, SRD Cohort 6: TAK-510 Dose 6 | Part 1, SRD Cohort 7: TAK-510 Dose 7 | Part 1, SRD Cohort 8: TAK-510 Dose 8 | Part 1, SRD Cohort 9: TAK-510 Dose 9 | Part 1, SRD Cohort 10: TAK-510 Dose 10 | Part 1, SRD Cohort 11: TAK-510 Dose 11 | Part 2, MRD 12 to 15 Cohorts: Pooled Placebo | Part 2, MRD Cohort 12: Dose 1A | Part 2, MRD Cohort 13: Dose 2A | Part 2, MRD Cohort 14: Dose 3A | Part 2, MRD Cohort 15: Dose 4A
Number analyzed (Participants) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Participants
  ADA Titer Low | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  ADA Titer High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Part 3: Number of ADA Positive Participants Based on Low or High ADA Titer
Description: The high ADA titer was defined as participant who has at least 1 post-baseline ADA titer >16 and low ADA titer was defined as participant whose postbaseline ADA titers are all <=16. Sponsor decided not to conduct Part 3 after comprehensive review of available data. No participants were enrolled in Part 3 of the study. Hence, no data collection and assessment were done in Part 3.
Time Frame: Part 3: From the first dose of study drug up to Day 29
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Parts 1 and 2, Cmax: Maximum Observed Plasma Concentration for TAK-510
Description: Due to confidentiality reasons and chances of exposing the doses for TAK-510, the data for this pharmacokinetic outcome measure was not reported.
Time Frame: Part 1, Day 1: pre-dose and at multiple time points (up to 96 hours) post-dose; Part 2, Day 1: pre-dose and at multiple time points (up to 24 hours) post-dose
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Part 1, AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-510
Description: as for outcome 13
Time Frame: Part 1, Day 1: pre-dose and at multiple time points (up to 96 hours) post-dose
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Part 1, AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-510
Description: as for outcome 13
Time Frame: Part 1, Day 1: pre-dose and at multiple time points (up to 96 hours) post-dose
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Parts 1 and 2, Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-510
Description: as for outcome 13
Time Frame: as for outcome 13
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Part 1, T1/2z: Terminal Disposition Phase Half-life for TAK-510
Description: as for outcome 13
Time Frame: Part 1, Day 1: pre-dose and at multiple time points (up to 96 hours) post-dose
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Part 1, CL/F: Apparent Clearance After Extravascular Administration for TAK-510
Description: as for outcome 13
Time Frame: Part 1, Day 1: pre-dose and at multiple time points (up to 96 hours) post-dose
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Part 1, Vz/F: Apparent Volume of Distribution During the Terminal Disposition Phase After Extravascular Administration for TAK-510
Description: as for outcome 13
Time Frame: Part 1, Day 1: pre-dose and at multiple time points (up to 96 hours) post-dose
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Part 2, AUCτ: Area Under the Plasma Concentration-time Curve Over a Dosing Interval for TAK-510
Description: as for outcome 13
Time Frame: Part 2, Day 1: pre-dose and at multiple time points (up to 24 hours) post-dose
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Part 2, AUCτss: Area Under the Plasma Concentration-time Curve Over a Dosing Interval at Steady State for TAK-510
Description: as for outcome 13
Time Frame: Part 2, Day 5: pre-dose and at multiple time points (up to 96 hours) post-dose
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Part 2, Cmaxss: Maximum Observed Plasma Concentration at Steady State for TAK-510
Description: as for outcome 13
Time Frame: Part 2, Day 5: pre-dose and at multiple time points (up to 96 hours) post-dose
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Part 2, Tmaxss: Time to Reach the Maximum Observed Plasma Concentration at Steady State for TAK-510
Description: as for outcome 13
Time Frame: Part 2, Day 5: pre-dose and at multiple time points (up to 96 hours) post-dose
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Part 2, T1/2z: Terminal Disposition Phase Half-life at Steady State for TAK-510
Description: as for outcome 13
Time Frame: Part 2, Day 5: pre-dose and at multiple time points (up to 96 hours) post-dose
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Part 2, CL/F: Apparent Clearance After Extravascular Administration at Steady State for TAK-510
Description: as for outcome 13
Time Frame: Part 2, Day 5: pre-dose and at multiple time points (up to 96 hours) post-dose
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Part 2, Vz/F: Apparent Volume of Distribution During the Terminal Disposition Phase After Extravascular Administration at Steady State for TAK-510
Description: as for outcome 13
Time Frame: Part 2, Day 5: pre-dose and at multiple time points (up to 96 hours) post-dose
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Part 2, Ctrough: Observed Plasma Concentration at the End of a Dosing Interval at Steady State for TAK-510
Description: as for outcome 13
Time Frame: Part 2, Day 5: pre-dose and at multiple time points (up to 96 hours) post-dose
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Part 2, Rac (AUC): Accumulation Ratio Based on AUCτ at Steady State for TAK-510
Description: as for outcome 13
Time Frame: Part 2, Day 5: pre-dose and at multiple time points (up to 96 hours) post-dose
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Part 2, Rac (Cmax): Accumulation Ratio Based on Cmax at Steady State for TAK-510
Description: as for outcome 13
Time Frame: Part 2, Day 5: pre-dose and at multiple time points (up to 96 hours) post-dose
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Parts 1 and 2, Aet: Amount of Drug Excreted in Urine From Time 0 to Time t for TAK-510
Description: as for outcome 13
Time Frame: Parts 1 and 2, Day 1: pre-dose and at multiple time points (up to 24 hours) post-dose
Reporting Status: Not Posted

31. Other Pre Specified Outcome: Parts 1 and 2, Aet1-t2: Amount of Drug Excreted in Urine From Time 1 to Time 2 for TAK-510
Description: as for outcome 13
Time Frame: Part 1, Day 1: pre-dose and at multiple time points (up to 24 hours) post-dose; Part 2, Days 1 and 5: pre-dose and at multiple time points (up to 24 hours) post-dose
Reporting Status: Not Posted

32. Other Pre Specified Outcome: Part 2, Aeτ: Amount of Drug Excreted in Urine During a Dosing Interval (Tau) at Steady State for TAK-510
Description: as for outcome 13
Time Frame: Part 2, Day 5: pre-dose and at multiple time points (up to 24 hours) post-dose
Reporting Status: Not Posted

33. Other Pre Specified Outcome: Parts 1 and 2, fe,t: Fraction of Administered Dose of Drug Excreted From Urine From Time 0 to Time t for TAK-510
Description: as for outcome 13
Time Frame: as for outcome 31
Reporting Status: Not Posted

34. Other Pre Specified Outcome: Parts 1 and 2, CLR: Renal Clearance for TAK-510
Description: as for outcome 13
Time Frame: as for outcome 31
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: TEAEs are AEs that started after the first dose of study drug until 30 days after last dose in Parts 1 and 2 (SRD Cohorts: up to Day 31, MRD Cohorts: up to Day 35)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- Part 2, MRD Cohort: Dose 1A: TAK-510 Dose 1A, injection, subcutaneously from Days 1 to 5. The dose of TAK-510 was based on safety, tolerability, and available PK data from SRD Part 1.
Arm/Group | Part 1, SRD Cohorts 1 to 11: Pooled Placebo | Part 1, SRD Cohort 1: TAK-510 Dose 1 | Part 1, SRD Cohort 2: TAK-510 Dose 2 | Part 1, SRD Cohort 3: TAK-510 Dose 3 | Part 1, SRD Cohort 4: TAK-510 Dose 4 | Part 1, SRD Cohort 5: TAK-510 Dose 5 | Part 1, SRD Cohort 6: TAK-510 Dose 6 | Part 1, SRD Cohort 7: TAK-510 Dose 7 | Part 1, SRD Cohort 8: TAK-510 Dose 8 | Part 1, SRD Cohort 9: TAK-510 Dose 9 | Part 1, SRD Cohort 10: TAK-510 Dose 10 | Part 1, SRD Cohort 11: TAK-510 Dose 11 | Part 2, MRD 12 to 15 Cohorts: Pooled Placebo | Part 2, MRD Cohort: Dose 1A | Part 2, MRD Cohort 13: Dose 2A | Part 2, MRD Cohort 14: Dose 3A | Part 2, MRD Cohort 15: Dose 4A
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/6 | 0/6 | 0/6 | 0/7 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/8 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/6 | 0/6 | 0/6 | 0/7 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/8 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 9/23 | 1/6 | 3/6 | 3/6 | 4/7 | 6/6 | 6/6 | 4/6 | 6/6 | 4/6 | 6/6 | 6/6 | 5/8 | 7/8 | 3/6 | 6/6 | 5/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1, SRD Cohorts 1 to 11: Pooled Placebo (N=23) | Part 1, SRD Cohort 1: TAK-510 Dose 1 (N=6) | Part 1, SRD Cohort 2: TAK-510 Dose 2 (N=6) | Part 1, SRD Cohort 3: TAK-510 Dose 3 (N=6) | Part 1, SRD Cohort 4: TAK-510 Dose 4 (N=7) | Part 1, SRD Cohort 5: TAK-510 Dose 5 (N=6) | Part 1, SRD Cohort 6: TAK-510 Dose 6 (N=6) | Part 1, SRD Cohort 7: TAK-510 Dose 7 (N=6) | Part 1, SRD Cohort 8: TAK-510 Dose 8 (N=6) | Part 1, SRD Cohort 9: TAK-510 Dose 9 (N=6) | Part 1, SRD Cohort 10: TAK-510 Dose 10 (N=6) | Part 1, SRD Cohort 11: TAK-510 Dose 11 (N=6) | Part 2, MRD 12 to 15 Cohorts: Pooled Placebo (N=8) | Part 2, MRD Cohort: Dose 1A (N=8) | Part 2, MRD Cohort 13: Dose 2A (N=6) | Part 2, MRD Cohort 14: Dose 3A (N=6) | Part 2, MRD Cohort 15: Dose 4A (N=6)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Arrhythmia supraventricular (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Blood pressure diastolic increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0 | 2 | 2 | 2 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram ST segment depression (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gingival discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Medical device site dermatitis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3 | 4 | 4 | 0 | 3 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 4
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 3 | 5 | 0 | 0 | 1 | 3 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scrotal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 5 | 0 | 3 | 2 | 4 | 5 | 5 | 4 | 6 | 4 | 6 | 2 | 2 | 6 | 2 | 6 | 5
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion

DOCUMENTS (2):
  • Study Protocol (2022-04-21): https://cdn.clinicaltrials.gov/large-docs/22/NCT04731922/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-31): https://cdn.clinicaltrials.gov/large-docs/22/NCT04731922/SAP_001.pdf